CLINICAL TRIAL: NCT05429710
Title: Immunohistochemical Expression of SOX2 and PD-L1 as Valuable Prognostic Markers in Urinary Bladder Carcinoma
Brief Title: SOX2 & PDL1 Expression on Urinary Bladder Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Salah, assisstant lecturer, Sohag University
Other Study IDs: Soh-med-22-06-13
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Urinary Bladder Neoplasm
Keywords: SOX2, PDL1, prgnosis, urinary bladder carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bladder carcinoma (BC) is the 13th leading cause of cancer mortality worldwide . In Egypt, BC is the third common malignant tumor. Its incidence is 8.7% of all malignant tumors in both sexes with more predominance in males as reported by National Cancer Registry with more expected cases in the future.

There are different histological variants of BC which show different phenotypic, biological and prognostic impacts. The most common histological type of BC is urothelial carcinoma which constitutes about 90% of all bladder cancers. Squamous cell carcinoma, adenocarcinoma and other rare types represent the remaining 10%.

Carcinoma of the bladder is considered a heterogeneous stem cell tumor with increasing morbidity and death rates if it is not treated properly. The presence of cancer stem cells (CSCs) is associated with tumor progression, recurrence, metastasis, and resistance to conventional chemotherapy and makes complete elimination of the tumor difficult. Successes in treatment plans need more understanding of the CSCs population and their molecular biology.

The most important items of CSCs regulatory core are transcription factors such as OCT4, SOX-2, and Nanog. They play an important role in the regulatory network for maintaining the 'stemness' state of stem cells.

SOX2 (short for Sex determing Region Y - box 2), a High Mobility Group (HMG) domain transcription factor is member of the SRY-related HMG-box (SOX) family of transcription factors involved in the pluripotency, self-reappearance and differentiation of embryonic stem cell.

Cancer immunotherapy starts with a proper understanding of tumor immuno-biology. Study of the tumor microenvironment revealed the importance of immune checkpoints in facilitating tumor immunological escape, leading to the development of multiple novel therapeutics targeting the PD-1/PD-L1 (programmed cell death protein 1, "CD279" programmed death ligand 1, "CD274") immune checkpoints. And recently the expression levels of PD-L1 are closely associated with CSCs immune escape.

PD-1 is a T-cell immune inhibitory checkpoint that inhibit T-cell activation and contributes to the immunosuppressive tumor microenvironment. PD-1 is also expressed on activated B cells and natural killer cells. PD-1 is activated by binding to its ligand; PD-L1, which is a type I trans-membrane glycoprotein. Many cell types express PD-L1, including placenta, vascular endothelium, hepatocytes and mesenchymal stem cells, also B cells, T cells, dendritic cells, macrophages, and mast cells.

PD-L1 is considered to be a co-inhibitory factor of the immune response, it can combine with PD-1 to reduce the proliferation of PD-1 positive cells, inhibit their cytokine secretion and induce apoptosis. PD-L1 also plays an important prognostic and predictive value in various malignancies where it can attenuate the host immune response to tumor cells.

However, little is known about the role of PD-L1 and its relation to SOX2 in urinary bladder carcinoma including its different histopathological variants. In this study, the main objective is to evaluate the immunohistochemical expression of PD-L1 to CSCs marker (SOX2) in urinary bladder carcinoma as a prognostic factor and search for new prospective targeted cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with urinary bladder carcinoma.
* Specimen with submitted muscle layer

Exclusion Criteria:

* Patients with insufficient clinical data.
* Patients with recurrence of the primary tumor.
* Specimens with extensive necrosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Formaline fixed and paraffine embedded urinary bladder tissue block from 60 patient
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Immunohistochemical Expression of SOX2 and PD-L1 as valuable prognostic markers in Urinary Bladder Carcinoma | one or two days after staining sections with the markers
  To evaluate the expression of SOX2 and PD-L1 in urinary bladder carcinomas

CONTACTS AND LOCATIONS:
Overall Officials: alaa MS elmaghraby, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: Undecided